CLINICAL TRIAL: NCT01458691
Title: Intra-articular Injection of Allogeneic PRP for Adhesive Capsulitis
Brief Title: Intra-articular Injection of Allogeneic Platelet Rich Plasma (PRP) for Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Associate Professor, SMG-SNU Boramae Medical Center, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM-11-02
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2015-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid group (Active Comparator): Triamcinolone injection group
  Interventions: Procedure: Steroid injection into the glenohumeral joint
- PRP group (Experimental): Allogeneic PRP injection group
  Interventions: Procedure: Allogeneic PRP injection into the glenohumeral joint

INTERVENTIONS:
Procedure: Steroid injection into the glenohumeral joint — * Group: Steroid
  * Total volume of injection drugs: 4ml(1ml of triamcinolone acetonide 40mg/ml + 3ml of 2% lidocaine)
  * The number of injections : only once during the study period
  * Injection site : glenohumeral joint
  * Material : 25-gauze spinal needle
  * The intra-articular injections were performed using ultrasonographic guidance.
  Arms: Steroid group
Procedure: Allogeneic PRP injection into the glenohumeral joint — * Group: Allogeneic PRP
  * Total volume of injection drugs: 4ml
  * The number of injections : only once during the study period
  * Injection site : glenohumeral joint
  * Material : 25-gauze spinal needle
  * The intra-articular injections were performed using ultrasonographic guidance.
  Arms: PRP group

SUMMARY:
The purpose of this study is to compare the efficacy of intra-articular allogenic Platelet Rich Plasma injection and steroid injection in the treatment of adhesive capsulitis of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age and older
2. Patients who have had pain at least for 12 months
3. limitation of both active and passive movements of the glenohumeral joint of ≥25% in at list 2 directions (abduction,flexion,external rotation,internal rotation), as compared with the contralateral shoulder in the scapular plane and in progressive degree of horizontal adduction

Exclusion Criteria:

1. Patients with concurrent bilateral shoulder pain
2. Patients with Diabetes mellitus
3. Patient with overt hypothyroidism or hyperthyroidism
4. Patients who received any drug by intra-articular injection for treatment within 6 months prior to this enrollment.
5. Patients who have a history of shoulder trauma including dislocation- subluxation- and fracture- breast cancer- or surgery around shoulder- neck and upper back
6. Patients with neurological deficit
7. Patients who have a History of allergic adverse reactions to corticosteroid
8. Patients with secondary adhesive capsulitis
9. Patients with systemic inflammatory disease including rheumatoid arthritis
10. Patients with degenerative arthritis, infectious arthritis of shoulder joint
11. Patients who have a history of shoulder trauma including dislocation, fracture
12. Patients taking anticoagulants
13. Patients who have a full-thickness rotator cuff tear
14. Patients who are difficulty participating in data collection due to communication problem and serious mental illness
15. Pregnant women or lactating mothers
16. Patients with cerebrovascular accident
17. Patients with symptomatic cervical spine disorders
18. Patients with serious condition which can affect this study such as severe cardiovascular diseases- renal diseases- liver diseases- endocrine diseases- and cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-10-20 (Actual)

PRIMARY OUTCOMES:
SPADI(Shoulder Pain and Disability Index)Score | Postinjection 1month
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.
Safety determined with symptoms & signs of infection and immune response and adverse events evaluated with NCI-CTCAE v3.0 | Postinjection 1month
  Presence of general symptoms or signs associated with infection and immune response, such as rash, pruritus, fever, chills, urticaria, or dyspnea.
  Injection sites were examined to identify erythema, swelling, or abnormal discharge.
  Adverse events were categorised with use of the National Cancer Institute Common Terminology Criteria for Adverse Events scale, version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Jo, M.D., Ph.D, Principal Investigator — Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea